CLINICAL TRIAL: NCT01214811
Title: Open Multi-centre Investigation to Evaluate Signs and Symptoms of Local Inflammation/Infection on Chronic Ulcers and Partial Thickness Burns When Using Mepilex Border Ag as an Anti-microbial Wound Dressing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxB Ag 01
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2011-12

CONDITIONS: Inflammation; Burns; Ulcers
Keywords: The change in signs of inflammation/local infection; To evaluate the comfort, conformability,; Pain during wear
MeSH Terms: conditions — Inflammation; Burns; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepilex Border Ag (Other): Non comparative study with one active arm - Mepilex Border Ag
  Interventions: Device: Mepilex Border Ag

INTERVENTIONS:
Device: Mepilex Border Ag — Mepilex Border Ag may be left in place for up to seven days, depending on the condition.

SUMMARY:
The purpose of this study is to evaluate the change in signs of inflammation/local infection when Mepilex Border Ag is used in normal clinical practice when used on chronic ulcers (venous leg, diabetic foot and pressure ulcers) and partial thickness burns in need* of topical antimicrobial treatment according to the physician.

DETAILED DESCRIPTION:
The investigation is designed as an open, non-controlled, post-marketing clinical follow-up. Subjects with chronic ulcers or partial thickness burns (including donor sites) at 2 sites will be included. Each subject with a chronic ulcer will be seen once a week for a maximum of 4 weeks or until desired treatment effect is obtained, whichever occurs earlier. Each subject with a partial thickness burn/donor site will be followed once a week for a maximum of 3 weeks or until desired treatment effect is obtained, whichever occurs earlier. All dressing changes will be done according to clinical routine practices and will follow IFU (instruction for use)

ELIGIBILITY:
Inclusion Criteria:

* Subject with a chronic ulcer (venous leg, diabetic foot and pressure ulcers) or a partial thickness burn where an antimicrobial action is indicated* as judged by the investigator
* Male or female, 18 years and above, both in- and out-patients
* Signed Informed Consent Form

Exclusion Criteria:

* Wound size equal to or above 9.5x15cm for the wound/burn to be included in the investigation
* Subject not expected to follow the investigation procedures
* TBSA > 10% (partial thickness burns only)
* HbA1C value > 7.2. (To be measured if BMI > 30)
* Pregnant and breastfeeding women
* Pressure ulcers deeper than stage 3
* Deep pressure ulcers in need of a filler
* Subjects with known sensitivity to silver or any other dressing materials
* Subjects receiving radiation treatment or examinations e.g. X-ray, ultrasound, diathermy or Magnetic Resonance Imaging
* Subjects using oxidising agents such as hypochlorite solutions or hydrogen peroxide
* Subjects previously included in this investigation
* Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Latenser, MD, Principal Investigator — UI burn Treatment Center,200 Hawkings Dr 8JCP Iowa City
Locations (3):
- United States (3):
  - Institute for advanced wound care, Momtgomery, Alabama
  - Burn treatment center, Iowa City, Iowa
  - Center for Curative & Palliative Care, Calvary Hospital, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Mepilex Border Ag: Non comparative study with one active arm - Mepilex Border Ag
  Mepilex Border Ag : Mepilex Border Ag may be left in place for up to seven days, depending on the condition.
Period: Overall Study
Arm/Group | Mepilex Border Ag
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Mepilex Border Ag
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Wound Are at Baseline
Time Frame: Baseline
Reporting Status: Not Posted

2. Primary Outcome: Wound Area at Visit 2
Description: At each visit the wound length and width is measured and calculated in cm2.
Time Frame: After one week
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Mepilex Border Ag
Number analyzed (Participants) | 27
cm2 | 43.0 (41.6)

ADVERSE EVENTS:
Arm/Group | Mepilex Border Ag
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No